CLINICAL TRIAL: NCT06745531
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: A Phase 3 Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS172-03-01
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hyperphosphatemia Patients on Hemodialysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TS-172 20~60 mg/day (Experimental)
  Interventions: Drug: TS-172 20~60 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-172 20~60 mg/day — oral administration of TS-172 20~60 mg/day
  Arms: TS-172 20~60 mg/day
Drug: Placebo — oral administration of placebo
  Arms: Placebo

SUMMARY:
A phase 3, randomized, placebo-controlled, double-blind study of TS-172 in hyperphosphatemia

ELIGIBILITY:
Inclusion Criteria:

1. Hyperphosphatemia patients (outpatients) with chronic kidney disease receiving hemodialysis (HD or HDF) 3 times a week for at least 12 weeks prior to Visit 1 (Week -4)
2. Patients aged >=18 years at the time of obtaining informed consent
3. Patients with a serum phosphorus concentration of >= 3.5 mg/dL and < 5.5 mg/dL at Visit 1 (Week -4)
4. Patients whose serum phosphorus concentration at Visit 3 (Week -2) or Visit 4 (Week -1) has increased by at least 1.0 mg/dL compared with the value at Visit 1 (Week -4) and is >= 5.5 mg/dL and < 10.0 mg/dL.

Exclusion Criteria:

1. Patients with confirmed serum intact PTH concentration >500 pg/mL from Visit 1 (Week -4) to Visit 5 (Week 0)
2. Patients with serum phosphorus concentration >= 10.0 mg/dL from Visit 2 (Week -3) to Visit 4 (Week -1)
3. Patients who have undergone previous parathyroid intervention (PTx, PEIT, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Achievement rate of the target serum phosphorus level | Week 8

SECONDARY OUTCOMES:
Change from baseline in serum concentration of phosphorus | Up to Week 8
Concentration of corrected serum calcium | Up to Week 8
Serum Ca × P product | Up to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan